CLINICAL TRIAL: NCT05302531
Title: Absorption of Antibiotics With High Oral Bioavailability in Short-bowel Syndrome : a Monocentric Pilot Study
Brief Title: Absorption of Antibiotics With High Oral Bioavailability in Short-bowel Syndrome
Acronym: GRAAL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Société Francophone Nutrition Clinique et Métabolisme (Other); FIlière des Maladies rares Abdomino-THOraciques (Unknown); Fresenius Kabi (Industry)
Responsible Party: Principal Investigator, MICHOT Niasha, Principal Investigator, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-001468-13
Record Dates: First submitted 2022-03-02; First posted 2022-03-31 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Short Bowel Syndrome; Infection, Bacterial
MeSH Terms: conditions — Short Bowel Syndrome; Bacterial Infections | interventions — Amoxicillin; Levofloxacin; Ofloxacin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Amoxicillin (Experimental): Each patient will receive the IV antibiotic required to treat the infection, and after the proper duration of the IV antibiotic is over, the patient will receive a few days of the oral version of the same antibiotic.
  Interventions: Drug: Amoxicillin
- Ofloxacin (Experimental): Each patient will receive the IV antibiotic required to treat the infection, and after the proper duration of the IV antibiotic is over, the patient will receive a few days of the oral version of the same antibiotic.
  Interventions: Drug: Ofloxacin
- Levofloxacin (Experimental): Each patient will receive the IV antibiotic required to treat the infection, and after the proper duration of the IV antibiotic is over, the patient will receive a few days of the oral version of the same antibiotic.
  Interventions: Drug: Levofloxacin
- Sulfamethoxazole trimethoprim (Experimental): Each patient will receive the IV antibiotic required to treat the infection, and after the proper duration of the IV antibiotic is over, the patient will receive a few days of the oral version of the same antibiotic.
  Interventions: Drug: Sulfamethoxazole trimethoprim

INTERVENTIONS:
Drug: Amoxicillin — Each patient will receive the proper antibiotic to treat the infection, first intravenously, then orally
  Arms: Amoxicillin
Drug: Levofloxacin — Each patient will receive the proper antibiotic to treat the infection, first intravenously, then orally
  Arms: Levofloxacin
Drug: Ofloxacin — Each patient will receive the proper antibiotic to treat the infection, first intravenously, then orally
  Arms: Ofloxacin
Drug: Sulfamethoxazole trimethoprim — Each patient will receive the proper antibiotic to treat the infection, first intravenously, then orally
  Arms: Sulfamethoxazole trimethoprim

SUMMARY:
The purpose of this study is to assess the drug absorption of oral antibiotics in patients with short bowel syndrome.

DETAILED DESCRIPTION:
When required, due to an infection, patients with short bowel syndrome will be treated with an intravenous antibiotic. The pharmacokinetic profile of that intravenous antibiotic will be determined. Once the full treatment with the intravenous antibiotic is over, the patient will be orally administered the same antibiotic, with determination of the oral pharmacokinetic profile, and both profiles will be compared, assessing the bioavailability of the oral antibiotic.

ELIGIBILITY:
Inclusion Criteria:

* Short bowel syndrome
* Treated for a documented infection with antibiogram by amoxicillin (+/- clavulanic acid)or ofloxacin or levofloxacin or sulfamethoxazole/trimethoprim
* Hospitalized in the Nutritional Assistant Unit or the Infectiology Unit of the Regional University Hospital of Nancy
* Affiliated to a social security system
* Having received an physical examination before entering study
* Having received full information regarding the study organization and having signed the informed consent

Exclusion Criteria:

* Patient at risk of worsening their oral absorption abilities during study
* Patient requiring dialysis
* Women of childbearing age without efficient birth control
* Allergy to any of the drugs tested
* Person concerned by Articles L. 1121-5, L. 1121-7 et L1121-8 of the Code of public health
* Person deprived of liberty or person undergoing psychiatric care pursuant to articles L. 3212-1 et L. 3213-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Assess the bioavailability of the oral antibiotic in patient with short bowel syndrome | Time -0.5 hours
  F (%)=(ASC PO)/(ASC IV) x (Dose IV)/(Dose PO)
Assess the bioavailability of the oral antibiotic in patient with short bowel syndrome | Time +0.5 hours
  F (%)=(ASC PO)/(ASC IV) x (Dose IV)/(Dose PO)
Assess the bioavailability of the oral antibiotic in patient with short bowel syndrome | Time +1 hour
  F (%)=(ASC PO)/(ASC IV) x (Dose IV)/(Dose PO)
Assess the bioavailability of the oral antibiotic in patient with short bowel syndrome | Time +1.5 hour
  F (%)=(ASC PO)/(ASC IV) x (Dose IV)/(Dose PO)
Assess the bioavailability of the oral antibiotic in patient with short bowel syndrome | Time +2 hours
  F (%)=(ASC PO)/(ASC IV) x (Dose IV)/(Dose PO)
Assess the bioavailability of the oral antibiotic in patient with short bowel syndrome | Time +4 hours
  F (%)=(ASC PO)/(ASC IV) x (Dose IV)/(Dose PO)
Assess the bioavailability of the oral antibiotic in patient with short bowel syndrome | Time +6 hours
  F (%)=(ASC PO)/(ASC IV) x (Dose IV)/(Dose PO)
Assess the bioavailability of the oral antibiotic in patient with short bowel syndrome | Time +8 hours
  F (%)=(ASC PO)/(ASC IV) x (Dose IV)/(Dose PO)

SECONDARY OUTCOMES:
Describe antibiotic absorption after oral administration in these patients | Time -0.5hour ; Time +0.5hour ; Time +1 hour ; Time+1.5 hour ; Time +2 hours ; Time+4 hours ; Time +6 hours ; Time + 8 hours
  Peak plasma concentration (Cmax) after oral intake
Describe antibiotic absorption after oral administration in these patients | Time -0.5hour ; Time +0.5hour ; Time +1 hour ; Time+1.5 hour ; Time +2 hours ; Time+4 hours ; Time +6 hours ; Time + 8 hours
  Peak plasma concentration time after oral intake (Tmax)
Describe antibiotic absorption after oral administration in these patients | Time -0.5hour ; Time +0.5hour ; Time +1 hour ; Time+1.5 hour ; Time +2 hours ; Time+4 hours ; Time +6 hours ; Time + 8 hours
  Area under the plasma concentration versus time curve (AUC)
Assess link between length of remaining bowel and antibiotic absorption | At inclusion
  Length of remaining bowel (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Niasha MICHOT, MD, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided
Depending on first results, this pilot study might be extended in a new multicenter study

REFERENCES:
- [Background] Scala-Bertola J, Rabiskova M, Lecompte T, Bonneaux F, Maincent P. Granules in the improvement of oral heparin bioavailability. Int J Pharm. 2009 Jun 5;374(1-2):12-6. doi: 10.1016/j.ijpharm.2009.02.020. Epub 2009 Mar 9. PMID 19446753
- [Background] American Gastroenterological Association. American Gastroenterological Association medical position statement: short bowel syndrome and intestinal transplantation. Gastroenterology. 2003 Apr;124(4):1105-10. doi: 10.1053/gast.2003.50139. No abstract available. PMID 12671903
- [Background] Pironi L, Arends J, Bozzetti F, Cuerda C, Gillanders L, Jeppesen PB, Joly F, Kelly D, Lal S, Staun M, Szczepanek K, Van Gossum A, Wanten G, Schneider SM; Home Artificial Nutrition & Chronic Intestinal Failure Special Interest Group of ESPEN. ESPEN guidelines on chronic intestinal failure in adults. Clin Nutr. 2016 Apr;35(2):247-307. doi: 10.1016/j.clnu.2016.01.020. Epub 2016 Feb 8. PMID 26944585
- [Background] Gupta A, Mehta Y, Juneja R, Trehan N. The effect of cannula material on the incidence of peripheral venous thrombophlebitis. Anaesthesia. 2007 Nov;62(11):1139-42. doi: 10.1111/j.1365-2044.2007.05180.x. PMID 17924895
- [Background] Maki DG, Kluger DM, Crnich CJ. The risk of bloodstream infection in adults with different intravascular devices: a systematic review of 200 published prospective studies. Mayo Clin Proc. 2006 Sep;81(9):1159-71. doi: 10.4065/81.9.1159. PMID 16970212
- [Result] Ward N. The impact of intestinal failure on oral drug absorption: a review. J Gastrointest Surg. 2010 Jun;14(6):1045-51. doi: 10.1007/s11605-009-1151-9. Epub 2010 Jan 22. PMID 20094812
- [Result] Vance-Bryan K, Guay DR, Rotschafer JC. Clinical pharmacokinetics of ciprofloxacin. Clin Pharmacokinet. 1990 Dec;19(6):434-61. doi: 10.2165/00003088-199019060-00003. PMID 2292168
- [Result] Lamp KC, Bailey EM, Rybak MJ. Ofloxacin clinical pharmacokinetics. Clin Pharmacokinet. 1992 Jan;22(1):32-46. doi: 10.2165/00003088-199222010-00004. PMID 1559306
- [Result] Barr WH, Zola EM, Candler EL, Hwang SM, Tendolkar AV, Shamburek R, Parker B, Hilty MD. Differential absorption of amoxicillin from the human small and large intestine. Clin Pharmacol Ther. 1994 Sep;56(3):279-85. doi: 10.1038/clpt.1994.138. PMID 7924123
- [Result] Severijnen R, Bayat N, Bakker H, Tolboom J, Bongaerts G. Enteral drug absorption in patients with short small bowel : a review. Clin Pharmacokinet. 2004;43(14):951-62. doi: 10.2165/00003088-200443140-00001. PMID 15530127
- [Result] Cheung YW, Barco S, Mathot RAA, van den Dool EJ, Stroobants AK, Serlie MJ, Middeldorp S, Coppens M. Pharmacokinetics of dabigatran etexilate and rivaroxaban in patients with short bowel syndrome requiring parenteral nutrition: The PDER PAN study. Thromb Res. 2017 Dec;160:76-82. doi: 10.1016/j.thromres.2017.10.025. Epub 2017 Nov 4. PMID 29127863
- [Result] Faye E, Drouet L, De Raucourt E, Green A, Bal-Dit-Sollier C, Boudaoud L, Corcos O, Bergmann JF, Joly F, Lloret-Linares C. Absorption and efficacy of acetylsalicylic acid in patients with short bowel syndrome. Ann Pharmacother. 2014 Jun;48(6):705-10. doi: 10.1177/1060028014526700. Epub 2014 Mar 25. PMID 24667978
- [Result] Thielke J, Martin J, Weber FL, Schroeder TJ, Goretsky S, Hanto DW. Pharmacokinetics of tacrolimus and cyclosporine in short-bowel syndrome. Liver Transpl Surg. 1998 Sep;4(5):432-4. doi: 10.1002/lt.500040502. No abstract available. PMID 9724482
- [Result] Ueno T, Tanaka A, Hamanaka Y, Suzuki T. Serum drug concentrations after oral administration of paracetamol to patients with surgical resection of the gastrointestinal tract. Br J Clin Pharmacol. 1995 Mar;39(3):330-2. doi: 10.1111/j.1365-2125.1995.tb04457.x. PMID 7619677
- [Result] Menardi G, Guggenbichler JP. Bioavailability of oral antibiotics in children with short-bowel syndrome. J Pediatr Surg. 1984 Feb;19(1):84-6. doi: 10.1016/s0022-3468(84)80023-8. PMID 6699766